CLINICAL TRIAL: NCT03162705
Title: Prospective Molecular Profiling in Small Cell Lung Cancer
Brief Title: Molecular Profiling in Small Cell Lung Cancer
Acronym: MPSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Sun Yat-sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-BLK-001
Record Dates: First submitted 2017-05-05; First posted 2017-05-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Lung Neoplasms; Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol is to obtain tumor tissues and blood samples from patients with a confirmed histological diagnosis of Small cell lung cancer(SCLC) for molecular profiling.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is most invasive subtypes of lung cancer. After diagnosis, the SCLC patients without treatment often die in 2-4 months. SCLC is a highly heterogeneous malignant tumor, the previous treatment principle of the tumor is based on the traditional histopathology, which not provide accurate guidance for precise treatment. In recent years, breakthrough has been made in molecular classification of breast cancer, non-small cell lung cancer, gastrointestinal cancer and of the other tumor, but SCLC molecular classification has not yet reported.

In this prospective study, SCLC tissues and blood samples from extensive SCLC patients will be obtained and evaluated of molecular profiling. Eligible population includes: patients who have not undergone any treatment and diagnosed of extensive SCLC by immunohistochemistry(IHC). The purpose is to evaluate molecular profiling of SCLC patients who are sensitive or resistant to chemotherapy (Cisplatin+Etoposide). To compare molecular alterations of SCLC patients with different prognosis (Overall Survival, Progress Free Survival).

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 75 years old.
* Sexes Eligible for Study: All
* Diagnosed of SCLC by IHC, and divided into extensive stage.
* The ECOG (Eastern Cooperative Oncology Group, ECOG) PS(performance status，PS) Scale score is 0 or 1.
* At least one measurable lesions by CT scan.
* Expect to survive for at least three months.
* Peripheral blood routine and liver and kidney function meet the following criterion (blood draw 7 days before the treatment begins) :
* The White Blood Cell (WBC) is greater than the 3.0×10^9/L or neutrophils (ANC) more than 1.5 x10^9/L;
* Hemoglobin (HGB) is greater than 80 g/L.
* Platelet (PLT) is greater than 100×10^9/L.
* (AST/ALT): Aspartate aminotransferase/Alanine aminotransferase<3.0 times of normal range.
* Total bilirubin (TBIL) < 1.5 times of normal range.
* Creatinine (CREAT) < 1.5 times of normal range.
* Female or male patients must adopt effective birth control measures.
* Informed consent forms provided. Patients must meet each of the above criteria.

Exclusion Criteria:

* Other pathological types of tumors ,rather than small cell lung cancer.
* Incorporating other tumors in the early diagnosis;
* Patients who have received chemotherapy, radiotherapy or any other anti-cancer treatment.
* Patients that known to be allergic to the drug components involved in the study;
* Patients with severe allergies or allergies;
* Pregnant or breastfeeding women;
* Patients with acute infection which is difficult to control;
* Drug abuse, substance abuse, long-term alcohol and AIDS(Acquired Immune Deficiency Syndrome) patients.

Candidates who meet each of the exclusion criteria will not included in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have been histologically diagnosed of small cell lung cancer and evaluated with extensive stage.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | Five years
  OS is defined as time duration from randomization until the date of death from any cause. If the participants who had survived after the end of the study, or loss of follow-up, their last time of contact is defined as a deadline.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Five years
  PFS is defined as time duration from randomization until the date of SD(Stable Disease) or PD(Progressed Disease) evaluated by WHO RECIST (World Health Organization Response Evaluation Criteria in Solid Tumors， Edition1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Linlang Guo, Principal Investigator — ZhuJiang Hostipal
Locations (1):
- Zhujiang Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lyu Q, Zhu W, Wei T, Ding W, Cao M, Wang Q, Guo L, Luo P, Zhang J. High mutations in fatty acid metabolism contribute to a better prognosis of small-cell lung cancer patients treated with chemotherapy. Cancer Med. 2021 Nov;10(21):7863-7876. doi: 10.1002/cam4.4290. Epub 2021 Sep 26. PMID 34564955